CLINICAL TRIAL: NCT00179062
Title: Effects of Risperidone and Olanzapine on Weight Gain, Physical Health, and Outcome in a Community Sample of Severity and Persistently Ill Patients
Brief Title: Effects of Risperidone and Olanzapine on Patients With Schizophrenia, Schizoaffective Disorder, Major Depression or Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Herbert Meltzer, M.D. - principal investigator, Vanderbilt Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 990472
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Depressive Disorder, Major; Bipolar Disorder
Keywords: major depression with psychotic features; bipolar disorder with psychotic features
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: olanzapine versus risperidone
- 2 (Active Comparator)
  Interventions: Drug: olanzapine versus risperidone

INTERVENTIONS:
Drug: olanzapine versus risperidone — Participants are to be randomized to olanzapine or risperidone. Antipsychotic medication will be given as per package insert daily for the twelve month duration of the trial.

SUMMARY:
This twelve month, open-label study considers the effect of Risperdal (risperidone) versus Zyprexa (olanzapine) on weight gain, physical health, and outcome in a population of those diagnosed with schizophrenia, schizoaffective disorder, major depression or bipolar disorder with psychotic features. This study evaluates symptom response as well as general health indicators such as body mass index, glucose, prolactin, and cholesterol levels at baseline, month (M)1, M3, M6 and M12.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for participation in the current research study.

1. Subjects will be males and females between 18-60 years of age
2. Subjects will have a definite diagnosis by DSM-IV criteria of schizophrenia, schizoaffective disorder, bipolar disorder or major depression with psychotic symptoms.
3. Subjects may be outpatients or inpatients at the time of entry. They will continue in the study if hospitalization should occur.
4. The subjects or their legal guardian must sign the informed consent form.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from consideration for the current research project.

1. Subjects will be excluded if they have a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis other than schizophrenia, schizoaffective disorder, bipolar disorder or depression with psychotic features; however, a concurrent diagnosis of post-traumatic stress disorder, which does not account for the subjects's psychosis is acceptable..
2. Subject has received continuous treatment of olanzapine or risperidone in the last two months.
3. Subjects receiving continuous treatment with olanzapine or risperidone in the last two months prior to entering the study will be excluded. This means the subject cannot have actually taken olanzapine or risperidone daily for more than four weeks prior to enrollment. There must be a gap of at least two days of not taking medication during that period. The dose for olanzapine cannot exceed 10 mg /day, the dose for risperidone 2 mg/day. The last day of exposure of any kind should be at least seven days before baseline.
4. Subject has been diagnosed as treatment refractory.
5. Subjects unable to speak or read the English language.
6. Subjects with a DSM-IV diagnosis of substance dependence within three months prior to selection. Occasional abuse (defined as bingeing no more than once per week) will not preclude entry.
7. Subjects with a documented disease of the central nervous system, including but not limited to stroke, tumor, Parkinson's disease, Alzheimer's disease, Huntington's disease, seizure disorder requiring anticonvulsants, history of brain trauma resulting in documented impairment, chronic infection, neurosyphilis.
8. Subjects with hepatic, renal, atherosclerotic heart disease, arrhythmias or gastrointestinal disease of sufficient degree to interfere with the excretion, absorption, and/or metabolism of trial medication.
9. Subjects with clinical signs of liver disease should be excluded.
10. Subjects with acute (e.g. infection), unstable (e.g. labile hypertension, unstable angina), significant, or untreated medical illness; patients with diastolic blood pressure > 95 mmHg at screening should be treated and stabilized before randomization.
11. Subjects with narrow angle glaucoma, chronic urinary retention and/or clinically significant prostatic hypertrophy, paralytic ileus or related conditions, which in the opinion of the investigator may be exacerbated by the anticholinergic effects of olanzapine.
12. Subjects with a known eating disorder
13. Female subjects who are pregnant or breast-feeding
14. Subjects who are being treated with a depot neuroleptic within one treatment cycle of the beginning of the washout period.
15. Subjects with a history of neuroleptic malignant syndrome.
16. Subjects with a high-risk for suicide.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2000-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the main and interactional effects of risperidone and olanzapine on body mass index (BMI), other measures of obesity, and other health-related factors, including total cholesterol, lipid panels, blood glucose, glycohemoglobin, and prolactin | twelve months

SECONDARY OUTCOMES:
Determine primary drug treatment effects and the relationships between change in BMI (body mass index), the biological measures listed above, and clinical outcomes including several domains of functioning. | twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Y Meltzer, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Psychiatric Hospital at Vanderbilt, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Meltzer HY, Bonaccorso S, Bobo WV, Chen Y, Jayathilake K. A 12-month randomized, open-label study of the metabolic effects of olanzapine and risperidone in psychotic patients: influence of valproic acid augmentation. J Clin Psychiatry. 2011 Dec;72(12):1602-10. doi: 10.4088/JCP.10m05997. Epub 2011 Jul 12. PMID 21813074